CLINICAL TRIAL: NCT01172002
Title: A Randomized Multicenter Trial Comparing Leflunomide and Azathioprine as Remission-Maintaining Treatment for Proliferative Lupus Glomerulonephritis.
Brief Title: Leflunomide Versus Azathioprine for Maintenance Therapy of Lupus Nephritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Changhai Hospital (Other); Shanghai 10th People's Hospital (Other); Shanghai Zhongshan Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); The First Affiliated Hospital of Soochow University (Other); Zhejiang University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Qilu Hospital of Shandong University (Other); AnHui ShengLi Hospital (Unknown); The First Affiliated Hospital of Bengbu Medical University (Other); The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: BaoChunde, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RenJiH-20100330
Record Dates: First submitted 2010-07-27; First posted 2010-07-29 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2010-08

CONDITIONS: Nephritis; Lupus
Keywords: Lupus Nephritis; Leflunomide; Azathioprine
MeSH Terms: conditions — Nephritis; Lupus Nephritis | interventions — Leflunomide; Azathioprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- leflunomide group (Experimental)
  Interventions: Drug: Leflunomide
- Azathioprine group (Active Comparator)
  Interventions: Drug: Azathioprine

INTERVENTIONS:
Drug: Leflunomide — Leflunomide, 20 mg/d, ORAL ,each day. Number of Cycles: until progression or unacceptable toxicity develops.
  Predonine, 10 mg/d, ORAL, each day. If extra renal flare occurs, the dose of predonine may be increased to 1mg/kg/day for not more than 2 weeks.
  Arms: leflunomide group
Drug: Azathioprine — Azathioprine,50-100 mg/d, ORAL ,each day . Number of Cycles: until progression or unacceptable toxicity develops.
  Predonine, 10 mg/d, ORAL, each day. If extra renal flare occurs, the dose of predonine may be increased to 1mg/kg/day for not more than 2 weeks.
  Arms: Azathioprine group

SUMMARY:
Leflunomide versus Azathioprine for Maintenance Therapy of Lupus Nephritis

DETAILED DESCRIPTION:
Proliferative glomerulonephritis is a common and severe manifestation of systemic lupus erythematosus (SLE) that usually requires intensive therapy with high doses of glucocorticosteroids and cytotoxic drugs, such as intravenous (IV) cyclophosphamide (CYC). The objective of this Trial is to compare leflunomide (LEF) and azathioprine (AZA), in terms of efficacy and toxicity, as remission-maintaining treatment of proliferative lupus glomerulonephritis, after a remission-inducing therapy with a short-course IV CYC regimen. The hypothesis of this trial is that LEF is non-inferior to AZA.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years
* Biopsy-proven proliferative lupus nephritis
* Disease activity, SLEDAI score ≥ 8 points
* Persistent proteinuria (≥ 1g/24h), with or without microscopic hematuria;
* Signed informed consent

Exclusion Criteria:

* Allergy to the LEF, CTX, AZA
* Recent treatment with high-dose glucocorticoids
* Weight <45kg
* Recent treatment with immunosuppressive drugs
* CNS( Central Nerve System) Lupus patients
* Hepatic failure patients
* Severely abnormal renal function or end-stage renal failure
* More exclusion criteria in the protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-03; Primary Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
lupus nephritis flare | two years

SECONDARY OUTCOMES:
24-hour proteinuria over time | two years
Serum albumin over time | two years
Number of extra renal flare | two years
Cumulated glucocorticoid intake | two years

CONTACTS AND LOCATIONS:
Overall Officials: Bao Chun De, Principal Investigator — RenJi Hospital
Locations (1):
- RenJi Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Fu Q, Wu C, Dai M, Wang S, Xu J, Dai L, Li Z, He L, Zhu X, Sun L, Lu L, Bao C. Leflunomide versus azathioprine for maintenance therapy of lupus nephritis: a prospective, multicentre, randomised trial and long-term follow-up. Ann Rheum Dis. 2022 Nov;81(11):1549-1555. doi: 10.1136/ard-2022-222486. Epub 2022 Jul 4. PMID 35788493